CLINICAL TRIAL: NCT02598050
Title: NIH Explanatory/Developmental Research Grant Program: Preoperative Cognitive Screening in Older Surgical Patients: Feasibility and Utility for Predicting Morbidity
Brief Title: Preoperative Cognitive Screening in Older Surgical Patients Utility for Predicting Morbidity
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gregory J. Crosby, M.D., Physician, Brigham and Women's Hospital
Other Study IDs: 2014P002400
Record Dates: First submitted 2015-09-30; First posted 2015-11-05 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Cognitive Impairment
Keywords: postoperative health outcomes; older surgical patients
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — White blood cells and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- older surgical patients: Patients 65 years of age and older having lower extremity joint replacement surgery.
  Interventions: Other: No Interventions as this is a observational study

INTERVENTIONS:
Other: No Interventions as this is a observational study

SUMMARY:
The purpose of this work is to determine whether preoperative cognitive screening of patients over the age of 65 can be used as predictor of postoperative outcomes in patients undergoing lower extremity surgical procedures. This work is important as it may aid patients, families and physicians about the appropriateness of the surgical procedure and in providing resources to patients who are at the highest risk of adverse outcomes.

DETAILED DESCRIPTION:
The overriding hypothesis is that preoperative cognitive impairment is a risk factor for poor surgical outcomes in seniors and that preoperative screening is superior to standard or systematic clinical processes for identifying at-risk patients. The first objective is to assess the marginal benefit of structured preoperative cognitive screening relative to standard or systematic preoperative evaluation for identifying seniors with likely cognitive impairment. The second objective is to determine whether preoperative cognitive impairment predicts postoperative outcome. This project is designed as a prospective, single-center observational study. The cohort will consist of 250 consenting subjects ≥ 65 years of age who present to the BWH Weiner Center for Preoperative Evaluation (CPE) prior to elective lower extremity joint replacement surgery. These surgeries are selected because they are common in this age group, associated with significant morbidity, and along with dementia are considered a priority area (bone and joint conditions) by AHRQ. These ages are chosen as significant clinical data demonstrate increased cognitive impairment in community dwelling elders. Eligibility criteria include: patients ≥ 65 years of age with an ASA physical status of I-IV presenting for elective joint replacement. Exclusion criteria will include planned ICU admission postoperatively, uncorrected vision or hearing impairment (unable to see pictures or read or hear instructions); limited use of the dominant hand (limited ability to draw); and or inability to speak, read, or understand English. Study staff will use the CPE computerized scheduling system, which is updated continuously in real time and captures relevant information such as age and procedure, to identify potential subjects. When patients check in with the receptionist in the CPE for their appointment they will be notified that they (and their surrogate) may be eligible to participate in a study in the CPE involving patients over the age of 65. The receptionist will then provide them with a brochure about the study that includes information about the purpose of the study, the risks to the patient, and the potential benefits to society. The patient will then be asked if they are willing to speak with one of the study investigators and only those patients that agree to speak with a study investigator will be approached. Patients with known cognitive impairment will be included in the study to determine whether this information is included in the preoperative evaluation form. They will sign their own consent if they are capable and going to sign their surgical procedure consent. In the event that the patient is not capable of signing their own consent a surrogate will be asked to provide consent with assent from the patient. In our prior studies with similar patient populations less than 1% had documented cognitive impairment. The staff member will then describe the goals and risks of the study in a quiet room in the PATC and ask the patient (and their surrogate where appropriate) if they choose to participate. After all questions have been answered and the patient has the opportunity to read the consent form, written consent will be obtained by one of the study investigators. After obtaining consent, study staff will gain information about the patient's age and years of education. Study staff will administer standard instruments to assess health and functional status (basic and instrumental activities of daily living [ADLs and IADLs, respectively, and the WHODAS]). The World Health Organization Disability Scale 2.0 (WHODAS) is an alternative to the SF36 to measure physical health and disability.

In addition, patients will be asked if they've had a fall within the last 6 months, whether they've been evaluated for a change in memory or thinking, who accompanied them to their appointment, their employment status, and their living situation (alone, institutionalized, living with family members) in a patient survey. The study staff will also administer the MiniCog, a simple cognitive screening tool that takes just 2-4 min to complete and has little or no education, language, or race bias. In addition, the Animal Fluency Test will be administered, which is a short cognitive screen that takes one minute to complete. Other measures of cognitive impairment will be obtained by study staff through: documentation on the patient's standard preoperative form, patient or informant report of diagnosis or evaluation for cognitive impairment or memory concerns, and systematic medical record review.

During their routine preoperative blood draw the phlebotomist will be provided with three heparinized blood tube labeled with only the patient's study ID number that will be returned to the investigative team and processed within 30 minutes of the blood draw. Briefly, half of the sample would be spun down and plasma harvested and stored at -80 degrees C and when an adequate sample size obtained used to measure inflammatory cytokines by ELISA. The remainder of the sample will be divided into 1-ml aliquots and incubated at 37°C for 15 min with phosphate-buffered saline (PBS) (control), 100 ng/ml interleukin (IL)-6, 100 ng/ml IL-10, or a combination of 100 ng/mlIL-2 and 2 ng/ml granulocyte macrophage colony-stimulating factor, or 1g/ml lipopolysaccharide. Blood samples will be resuspended in 1.4 ml stabilizing buffer and incubated for 10 min at room temperature for fixation in PFA, cooled to 4C, and stored at 80C until further processing for flow cytometry to determine the immune response of the white blood cells to a ex-vivo immune challenge and whether these correlate with Mini-Cog score or the development of delirium.

Each enrolled patient will receive a business card listing the investigators' contact information and be advised to expect a follow up telephone call 6 months and 1 year after surgery to verify data elements and reassess functional outcome. Delirium will be assessed prospectively once per day on postoperative days 1, 2, and 3 by a trained study team member using the Confusion Assessment Method [CAM]. Delirium is most common on postoperative days 1-3 and the CAM is a well-validated measure of delirium in surgical patients. For functional status, the WHODAS will be administered 6-12 months postoperatively either by personnel in the surgeon's office as part of routine follow up or by study staff or by telephone. Investigators will also collect information on secondary outcomes including duration of PATC visit, presence of an advanced directive, whether they had surgical procedure, time to PACU discharge, discharge to place other than home (rehabilitation, skilled nursing facility), hospital length of stay (LOS), in hospital complications, perioperative variables including drugs administered, BIS, estimated blood loss, blood transfusions, fluid administered, blood pressure, oxygen saturation, 30-day reoperation or readmission rate, and 30-day and 1-year mortality. These outcomes are recorded in the medical record, the BWH Balanced Scorecard, an electronic database of all hospitalized patients that tabulates 31 elements of the hospital event, or the BWH Research Patient Database Enhanced Query. Data will also be confirmed by a follow up telephone interview. Thirty day and 1 year mortality will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* consenting patients ≥ 65 years of age
* undergoing upcoming elective lower joint replacement surgery

Exclusion Criteria:

* planned ICU admission postoperatively
* uncorrected vision or hearing impairment
* limited use of the dominant hand
* inability to speak, read, or understand English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This project is designed as a prospective, single-center observational study. The cohort will consist of 250 consenting subjects ≥ 65 years of age who present to the BWH Weiner Center for Preoperative Evaluation (CPE) prior to elective lower extremity joint replacement surgery. Eligibility criteria include: patients ≥ 65 years of age with an ASA physical status of I-IV presenting for elective joint replacement. Exclusion criteria will include planned ICU admission postoperatively, uncorrected vision or hearing impairment (unable to see pictures or read or hear instructions); limited use of the dominant hand (limited ability to draw); and or inability to speak, read, or understand English.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
CAM Score Postoperative Day 1-3 | Up to 3 days after surgery
  patient score on the Confusion Assessment Method and comprehensive chart review up to 1, 2, or 3 days after surgery

SECONDARY OUTCOMES:
Number of newly diagnosed health complications | up to 30 days after surgical procedure
  Newly diagnosed health complications up to 30 days after the surgical procedure including: Myocardial Infarction, CHF, Cardiac Arrest, Arrythmia, Pneumonia, PE, Reintubation, Stroke, Delirium, Coma>24h, deep wound infection,Superficial wound infection, Sepsis, Renal Failure, UTI, Reoperation, DVT, ICU admission,
Discharge location (Home vs. other than home) on the day of patient discharge from hospital | up to 30 days after the surgical procedure.
  day discharged to home or other than home
Number of days between surgical procedure and day of discharge | up to 30 days after surgical procedure
  number of days patient stayed in hospital following surgical procedure
30 day mortality | 30 days after surgical procedure
  patient mortality 30 days after surgical procedure
30 day re-operation or readmission | 30 days after surgical procedure
  patient readmission to the hospital or reoperation 30 days after surgical procedure
1 year mortality | 1 year after surgical procedure
  patient mortality 1 year after surgical procedure
Functional health outcome | 6 months-1 year after surgical procedure
  functional health outcome measured with the SF36 6 months to 1 year following the patient's surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Culley, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Weiner Center for Preoperative Evaluation, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT02598050/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT02598050/ICF_001.pdf